CLINICAL TRIAL: NCT02495194
Title: Effects of Horticultural Therapy on Asian Elderly' Mental Health: A Randomized Controlled Trial
Brief Title: Effects of Horticultural Therapy on Asian Elderly' Mental Health
Acronym: HTRCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: National Parks Board, Singapore (Other)
Responsible Party: Principal Investigator, Roger Ho Chun Man, Consultant Psychiatrist, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: B-15-016
Record Dates: First submitted 2015-06-24; First posted 2015-07-13 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Mood (Psychological Function)
Keywords: Promotion of psychological well-being; Horticultural therapy; Randomized Controlled Trial; Gardening; Elderly
MeSH Terms: interventions — Horticultural Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Horticultural Therapy (Experimental): 15 sessions of Horticultural Therapy program teaching the elderly about gardening techniques and for them to benefit from the therapeutic effects of the parks
  Interventions: Behavioral: Horticultural Therapy
- Waitlist Control Group (Other): Participants will receive the same horticultural therapy program at the end of the assessments
  Interventions: Behavioral: Horticultural Therapy

INTERVENTIONS:
Behavioral: Horticultural Therapy — The Horticultural Therapy intervention consists of 1 hour sessions weekly for first 3 months, followed by monthly session for the next 3 months. They will be taught on the basic gardening techniques such as sowing, weeding and fertilization during the hands-on sessions. They will also be taken on walks to the various parks to enjoy the therapeutic effect of the park greenery

SUMMARY:
The objective of this study is to determine whether horticultural therapy would improve the psychological well-being of the older adults. 70 healthy elderly were randomized into the active horticultural therapy or the waitlist control group. Sessions will be conducted weekly for 12 weeks, and monthly for 3 months. Participants would be assessed at 3 time-points: at the start, at 3-months and at 6-months.

It was hypothesized that as compared to the waitlist control group, participants in the active horticultural therapy will have (1) lower depression and anxiety symptomatology; (2) higher life satisfaction; (3) feel more socially connected; and (4) improved cognitive functioning.

DETAILED DESCRIPTION:
Participants Study participants are community-dwelling elderly.

Assessments Demographic data will be collected at the start. Psychological tests for depression, anxiety and psychological well-being as well as neuropsychological tests of cognitive functioning will be done at the start, at 3-months and at 6-months. Blood samples will also be collected at all three time points.

Intervention Sessions This is an intervention study with a waitlist control group design. The strength of this design is its experimental nature with randomization.

The Horticultural Therapy intervention is delivered by a trained practitioner at various locations and consists of 1 hour sessions weekly for first 3 months, followed by monthly session for the next 3 months. The extension of monthly sessions for 3 months is to determine sustainability and longer-term changes. The intervention is designed to cultivate an interest in gardening and promote relaxation. This will be achieved in stages, facilitated by trained volunteers and practitioners. The plant would be selected based on subjects' profiles e.g. familiarity, preference, safety and its maintenance would be followed up every fortnight. Park venues were selected based on patients profiles and park features e.g. familiarity, comfort under weather, safety.

The control group will be placed on a waiting list and only be contacted for assessments. They will receive intervention after the active treatment group at a later date.

The horticultural therapy is conducted solely for the purpose of this research.

ELIGIBILITY:
Inclusion criteria:

1. Community-living elderly aged between 60 to 85 years AND
2. able to provide informed consent AND
3. function independently AND
4. With a minimum score of 22 and above on the Montreal Cognitive Assessment.

Exclusion criteria:

1. Those who do not meet the above inclusion criteria (ie. Do not have a MCI diagnosis),
2. Does not have a minimum score of 22 and above on the Montreal Cognitive Assessment OR
3. Currently suffering from or have history of severe medical conditions e.g. cancer, stroke, Parkinson disease OR
4. History of severe psychiatric conditions e.g. schizophrenia, bipolar disorder OR
5. Dementia OR
6. Undergoing another therapy at the same time OR
7. Significant visual or hearing impairment OR
8. Marked upper and lower limb motor difficulties, which may affect their ability to participate in the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Zung Self-Rating Depression Scale (SDS) at 3-months and 6-months | baseline, 3-months, 6-months
  The SDS (Zung, 1965) is a 20-item quantitative measurement of symptoms of depression. Participants rate each item regarding how they felt during the week preceding using a 4-point scale that ranges from 1 (a little of the time) to 4 (most of the time). A total raw score computed by summing the scores on the individual items will be converted into a percentage (the SDS index); the higher the SDS index, the greater the severity of depressive symptoms. Several studies have established the SDS as a reliable and valid instrument for measuring depressive symptoms (Biggs et al., 1978; Gabrys and Peters, 1985; Agrell and Dehlin, 1989).
Change from baseline Zung Self-Rating Anxiety Scale (SAS) at 3-months and 6-months | baseline, 3-months, 6-months
  The SAS (Zung, 1971) will be used to measure anxiety of the participants in the preceding week. It is a 20-item self-report assessment designed to measure anxiety levels, based on cognitive, autonomic, motor and central nervous system symptoms. Each question is scored on a Likert-type scale of 1-4 (a little of the time) to (most of the time). Some questions are negatively worded to avoid the problem of set response. Overall assessment is done by total score. The total raw scores range from 20-80. The raw score then needs to be converted to an "Anxiety Index" score; the higher the SAS index, the greater the severity of depressive symptoms.
Change from baseline Ryff's Scales of Psychological Well-being at 3-months and 6-months | baseline, 3-months, 6-months
  The Ryff Scales of Psychological Well-Being (Ryff and Singer, 1998) is an 18-item questionnaire which reflects the six areas of psychological well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Respondents rate statements on a scale of 1 to 6, with 1 indicating strong disagreement and 6 indicating strong agreement.
Change from baseline Satisfaction with Life Scale (SWLS) at 3-months and 6-months | baseline, 3-months, 6-months
  Satisfaction with Life Scale (SWLS; Diener, Emmons, Larsen and Griffin, 1985) will be administered. SWLS is a 5-item scale designed to measure global cognitive judgments of one's life satisfaction (not a measure of either positive or negative affect). It is a psychometrically sound measure (Larson, Diener and Emmons, 1985) and has been validated in a geriatric population (Diener et al., 1985). Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 1 (strongly disagree) to 7 (strongly agree). Total scores were computed by summing the scores on the individual items and ranged from 5 to 35, with higher scores indicating higher level of satisfaction with life.
Change from baseline Friendship Scale (FS) at 3-months and 6-months | baseline, 3-months, 6-months
  Social connectedness scale will be measured using the Friendship Scale (Hawthorne, 2006). It is a 6-item questionnaire that measures both social isolation and social connectedness. Participants were asked to rate the frequency in which each statement describes them during the past four weeks on a 5-point Likert scale ranging from 0 (almost always) to 5 (not at all). Total scores were computed by summing the scores on the individual items and ranged from 0 to 24, with higher scores indicating higher level of social connectedness. The Friendship Scale was developed as a short, user-friendly, stand alone scale measuring perceived social isolation. It was validated with older adults with excellent internal structures, reliability and validity (Hawthorne, 2006; Hawthorne, 2008).
Change from baseline Interleukin 6 (IL-6) at 3-months and 6-months | baseline, 3-months, 6-months
  10ml of fasting blood will be collected using CPT tube
Change from baseline Interleukin-1 beta (IL-1β) at 3-months and 6-months | baseline, 3-months, 6-months
  10ml of fasting blood will be collected using CPT tube
Change from baseline C-reactive protein (CRP) at 3-months and 6-months | baseline, 3-months, 6-months
  10ml of fasting blood will be collected using CPT tube
Change from baseline Cortisol at 3-months and 6-months | baseline, 3-months, 6-months
  10ml of fasting blood will be collected using CPT tube
Change from baseline Brain-derived neurotrophic factor (BDNF) at 3-months and 6-months | baseline, 3-months, 6-months
  10ml of fasting blood will be collected using CPT tube
Change from baseline Dehydroepiandrosterone sulphate (DHEAS) at 3-months and 6-months | baseline, 3-months, 6-months
  10ml of fasting blood will be collected using CPT tube

SECONDARY OUTCOMES:
Change from baseline Montreal Cognitive Assessment (MoCA) at 3-months and 6-months | baseline, 3-months, 6-months
  Montreal Cognitive Assessment (MoCA) (Nasreddine, Phillips, Bedirian, Charbonneau, Whitehead, Collin, et al., 2005) will be administered by trained research assistants and/or research nurses as global measures of cognitive function.
Change from baseline Clinical Dementia Rating (CDR) at 3-months and 6-months | baseline, 3-months, 6-months
  Clinical Dementia Rating (CDR ) is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care.
Change from baseline Rey Auditory Verbal Learning Test (RAVLT) at 3-months and 6-months | baseline, 3-months, 6-months
  Rey Auditory Verbal Learning Test (RAVLT) evaluates declarative verbal learning and memory.
Change from baseline Digit Span Task at 3-months and 6-months | baseline, 3-months, 6-months
  Digit Span Task, which consists of a Digit Span Forward (DSF) and a Digit Span Backward (DSB) task is used to assess attention and verbal working memory.
Change from baseline Colour Trails Tests (CTT) at 3-months and 6-months | baseline, 3-months, 6-months
  Colour Trails Tests (CTT) 1 and 2 assesses sustained attention and sequencing.
Change from baseline Block Design at 3-months and 6-months | baseline, 3-months, 6-months
  Block Design is a subtest that is administered as part of several of the Wechsler Intelligence tests, and it primarily measures visual-spatial and organizational processing abilities, as well as non-verbal problem-solving skills.
Change from baseline Semantic Verbal Fluency at 3-months and 6-months | baseline, 3-months, 6-months
  Semantic Verbal Fluency taps lexical knowledge and semantic memory organization.
Change from Basic Health Screen (composite) at 3-months and 6-months | baseline, 3-months, 6-months
  Blood pressure, Pulse rate, Height and Weight will be measured

OTHER OUTCOMES:
Demographic questionnaire | Baseline
  Their social, demographic, and lifestyle data (i.e. how often they usually visit the parks or do gardening) will only be collected at baseline. This is the same for the participants' medical conditions.
Feedback questionnaire | Baseline
  Feedback questionnaire will be conducted to convey participants' subjective experience and thereby expanding our understanding of the impact of the horticultural therapy intervention. The survey will ask participants to identify what was the most helpful part of the class, what suggestions they have for improvement, and whether they had continued gardening and/or visiting the parks. This brief survey will only be administered once during the post-intervention assessment. Participants' responses will be informally tallied and listed in categories.

CONTACTS AND LOCATIONS:
Overall Officials: Roger CM Ho, FRCP, Principal Investigator — National University of Hospital
Locations (1):
- Training and Research Academy; Jurong Point Shopping Centre, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Aydemir C, Yalcin ES, Aksaray S, Kisa C, Yildirim SG, Uzbay T, Goka E. Brain-derived neurotrophic factor (BDNF) changes in the serum of depressed women. Prog Neuropsychopharmacol Biol Psychiatry. 2006 Sep 30;30(7):1256-60. doi: 10.1016/j.pnpbp.2006.03.025. Epub 2006 May 2. PMID 16647794
- [Background] Barnicle, T., & Midden, K. S. (2003). The effects of a horticulture activity program on the psychological well-being of older people in a long-term care facility. HortTechnology, 13(1), 81-85.
- [Background] Baune BT, Smith E, Reppermund S, Air T, Samaras K, Lux O, Brodaty H, Sachdev P, Trollor JN. Inflammatory biomarkers predict depressive, but not anxiety symptoms during aging: the prospective Sydney Memory and Aging Study. Psychoneuroendocrinology. 2012 Sep;37(9):1521-30. doi: 10.1016/j.psyneuen.2012.02.006. Epub 2012 Mar 9. PMID 22406002
- [Background] BOARD F, PERSKY H, HAMBURG DA. Psychological stress and endocrine functions; blood levels of adrenocortical and thyroid hormones in acutely disturbed patients. Psychosom Med. 1956 Jul-Aug;18(4):324-33. doi: 10.1097/00006842-195607000-00006. No abstract available. PMID 13350458
- [Background] Brunoni AR, Lopes M, Fregni F. A systematic review and meta-analysis of clinical studies on major depression and BDNF levels: implications for the role of neuroplasticity in depression. Int J Neuropsychopharmacol. 2008 Dec;11(8):1169-80. doi: 10.1017/S1461145708009309. Epub 2008 Aug 28. PMID 18752720
- [Background] Chu, C. M., & Simpson, R. (1994). Ecological public health: from vision to practice. Centre for Health Promotion, University of Toronto: ParticipACTION.
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486
- [Background] Gervasoni N, Aubry JM, Bondolfi G, Osiek C, Schwald M, Bertschy G, Karege F. Partial normalization of serum brain-derived neurotrophic factor in remitted patients after a major depressive episode. Neuropsychobiology. 2005;51(4):234-8. doi: 10.1159/000085725. Epub 2005 May 12. PMID 15897674
- [Background] GIBBONS JL. CORTISOL SECRETION RATE IN DEPRESSIVE ILLNESS. Arch Gen Psychiatry. 1964 Jun;10:572-5. doi: 10.1001/archpsyc.1964.01720240026004. No abstract available. PMID 14159257
- [Background] GIBBONS JL, McHUGH PR. Plasma cortisol in depressive illness. J Psychiatr Res. 1962 Sep;1:162-71. doi: 10.1016/0022-3956(62)90006-7. No abstract available. PMID 13947658
- [Background] Gonzalez MT, Hartig T, Patil GG, Martinsen EW, Kirkevold M. A prospective study of existential issues in therapeutic horticulture for clinical depression. Issues Ment Health Nurs. 2011;32(1):73-81. doi: 10.3109/01612840.2010.528168. PMID 21208054
- [Background] Gonzalez MT, Hartig T, Patil GG, Martinsen EW, Kirkevold M. Therapeutic horticulture in clinical depression: a prospective study of active components. J Adv Nurs. 2010 Sep;66(9):2002-13. doi: 10.1111/j.1365-2648.2010.05383.x. Epub 2010 Jul 2. PMID 20626473
- [Background] Grahn, P., & Stigsdotter, U. A. (2003). Landscape planning and stress. Urban forestry & urban greening, 2(1), 1-18.
- [Background] Hancock, T. (1999). Health care reform and reform for health: creating a health system for communities in the 21st century. Futures, 31(5), 417-436.
- [Background] Hartig, T., Evans, G. W., Jamner, L. D., Davis, D. S., & Gärling, T. (2003). Tracking restoration in natural and urban field settings. Journal of environmental psychology, 23(2), 109-123.
- [Background] Hayashi, N., Wada, T., Hirai, H., Miyake, T., Matsuura, Y., Shimizu, N., Kurooka, H. & Horiuchi, S. (2008). The effects of horticultural activity in a community garden on mood changes. Environmental Control in Biology, 46(4), 233-240.
- [Background] Henrich J, Heine SJ, Norenzayan A. Most people are not WEIRD. Nature. 2010 Jul 1;466(7302):29. doi: 10.1038/466029a. No abstract available. PMID 20595995
- [Background] Hiles SA, Baker AL, de Malmanche T, Attia J. A meta-analysis of differences in IL-6 and IL-10 between people with and without depression: exploring the causes of heterogeneity. Brain Behav Immun. 2012 Oct;26(7):1180-8. doi: 10.1016/j.bbi.2012.06.001. Epub 2012 Jun 9. PMID 22687336
- [Background] Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosom Med. 2009 Feb;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. Epub 2009 Feb 2. PMID 19188531
- [Background] Jeste DV, Alexopoulos GS, Bartels SJ, Cummings JL, Gallo JJ, Gottlieb GL, Halpain MC, Palmer BW, Patterson TL, Reynolds CF 3rd, Lebowitz BD. Consensus statement on the upcoming crisis in geriatric mental health: research agenda for the next 2 decades. Arch Gen Psychiatry. 1999 Sep;56(9):848-53. doi: 10.1001/archpsyc.56.9.848. PMID 12884891
- [Background] Kam, M. C., & Siu, A. M. (2010). Evaluation of a horticultural activity programme for persons with psychiatric illness. Hong Kong Journal of Occupational Therapy, 20(2), 80-86.
- [Background] Kamioka H, Tsutani K, Yamada M, Park H, Okuizumi H, Honda T, Okada S, Park SJ, Kitayuguchi J, Abe T, Handa S, Mutoh Y. Effectiveness of horticultural therapy: a systematic review of randomized controlled trials. Complement Ther Med. 2014 Oct;22(5):930-43. doi: 10.1016/j.ctim.2014.08.009. Epub 2014 Sep 1. PMID 25440385
- [Background] Karege F, Perret G, Bondolfi G, Schwald M, Bertschy G, Aubry JM. Decreased serum brain-derived neurotrophic factor levels in major depressed patients. Psychiatry Res. 2002 Mar 15;109(2):143-8. doi: 10.1016/s0165-1781(02)00005-7. PMID 11927139
- [Background] Kim YK, Lee HP, Won SD, Park EY, Lee HY, Lee BH, Lee SW, Yoon D, Han C, Kim DJ, Choi SH. Low plasma BDNF is associated with suicidal behavior in major depression. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jan 30;31(1):78-85. doi: 10.1016/j.pnpbp.2006.06.024. Epub 2006 Aug 10. PMID 16904252
- [Background] Lee BH, Kim H, Park SH, Kim YK. Decreased plasma BDNF level in depressive patients. J Affect Disord. 2007 Aug;101(1-3):239-44. doi: 10.1016/j.jad.2006.11.005. Epub 2006 Dec 13. PMID 17173978
- [Background] Kua EH. A community study of mental disorders in elderly Singaporean Chinese using the GMS-AGECAT package. Aust N Z J Psychiatry. 1992 Sep;26(3):502-6. doi: 10.3109/00048679209072077. PMID 1417639
- [Background] Kua E.H., Ko, S.M., Fones, C.S.L., & Tan S.L. (1997a). Epidemiology of depression in elderly Chinese living in Singapore. Journal of American Medical Association (Suppl), 13: 29-32.
- [Background] Liu Y, Ho RC, Mak A. Interleukin (IL)-6, tumour necrosis factor alpha (TNF-alpha) and soluble interleukin-2 receptors (sIL-2R) are elevated in patients with major depressive disorder: a meta-analysis and meta-regression. J Affect Disord. 2012 Aug;139(3):230-9. doi: 10.1016/j.jad.2011.08.003. Epub 2011 Aug 26. PMID 21872339
- [Background] Milligan C, Gatrell A, Bingley A. "Cultivating health": therapeutic landscapes and older people in northern England. Soc Sci Med. 2004 May;58(9):1781-93. doi: 10.1016/S0277-9536(03)00397-6. PMID 14990378
- [Background] Owen BM, Eccleston D, Ferrier IN, Young AH. Raised levels of plasma interleukin-1beta in major and postviral depression. Acta Psychiatr Scand. 2001 Mar;103(3):226-8. doi: 10.1034/j.1600-0447.2001.00162.x. PMID 11240580
- [Background] Sen S, Duman R, Sanacora G. Serum brain-derived neurotrophic factor, depression, and antidepressant medications: meta-analyses and implications. Biol Psychiatry. 2008 Sep 15;64(6):527-32. doi: 10.1016/j.biopsych.2008.05.005. Epub 2008 Jun 24. PMID 18571629
- [Background] Shimizu E, Hashimoto K, Okamura N, Koike K, Komatsu N, Kumakiri C, Nakazato M, Watanabe H, Shinoda N, Okada S, Iyo M. Alterations of serum levels of brain-derived neurotrophic factor (BDNF) in depressed patients with or without antidepressants. Biol Psychiatry. 2003 Jul 1;54(1):70-5. doi: 10.1016/s0006-3223(03)00181-1. PMID 12842310
- [Background] Thomas AJ, Davis S, Morris C, Jackson E, Harrison R, O'Brien JT. Increase in interleukin-1beta in late-life depression. Am J Psychiatry. 2005 Jan;162(1):175-7. doi: 10.1176/appi.ajp.162.1.175. PMID 15625217
- [Background] Tse MM. Therapeutic effects of an indoor gardening programme for older people living in nursing homes. J Clin Nurs. 2010 Apr;19(7-8):949-58. doi: 10.1111/j.1365-2702.2009.02803.x. PMID 20492039
- [Background] Valkanova V, Ebmeier KP, Allan CL. CRP, IL-6 and depression: a systematic review and meta-analysis of longitudinal studies. J Affect Disord. 2013 Sep 25;150(3):736-44. doi: 10.1016/j.jad.2013.06.004. Epub 2013 Jul 17. PMID 23870425
- [Derived] Chan HY, Ho RC, Mahendran R, Ng KS, Tam WW, Rawtaer I, Tan CH, Larbi A, Feng L, Sia A, Ng MK, Gan GL, Kua EH. Effects of horticultural therapy on elderly' health: protocol of a randomized controlled trial. BMC Geriatr. 2017 Aug 29;17(1):192. doi: 10.1186/s12877-017-0588-z. PMID 28851276